CLINICAL TRIAL: NCT00038389
Title: Phase I Study of Vioxx and Radiation Therapy for Brainstem Glioma
Brief Title: Study of Vioxx and Radiation Therapy for Brainstem Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unavailability of study drug.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID01-460
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Glioma; Brain Neoplasms
Keywords: Brain Stem Tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms; Brain Stem Neoplasms | interventions — rofecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vioxx MTD (Experimental)
  Interventions: Drug: Vioxx

INTERVENTIONS:
Drug: Vioxx — Starting dose for patients age 3-14 years 10.0 mg/1.73 m2 and for patients above 14 years of age 12.5 mg for 5 days per week for 6 weeks during radiation treatment, and 7 days per week for 6 months after radiation treatment.
  Other Names: Rofecoxib

SUMMARY:
It is of interest to determine whether COX-2 inhibitors given with radiation therapy can prolong the progression-free survival in brain stem glioma. Diffuse pontine brainstem gliomas are more common in children, but are also seen in adults. However, the use of commercially available COX-2 inhibitors has not been evaluated in the pediatric population and the proper dosing in pediatrics is unknown. Therefore a Phase I study will need to be conducted as a first step. Rofecoxib is an FDA approved COX-2 inhibitor for use in adults. This phase I study is designed to determine the maximum tolerated dose of Rofecoxib given concurrently with standard radiation therapy for diffuse pontine brainstem glioma.

DETAILED DESCRIPTION:
Rofecoxib is a non-steroidal anti-inflammatory drug.

Patients in this study will take a certain amount of rofecoxib by mouth either once or twice a day during treatment with radiation therapy. They will continue to take rofecoxib for 6 months after the end of radiation therapy. Different dose levels will be given to different patients based on a statistical dose escalation (increase) program run on a computer called the Continuous Reassessment Method. At least 3 patients will be treated on each dose level starting at the lowest level. All patients are required to fill out a medication diary, documenting the dose of rofecoxib they are taking and the time they take it.

Patients will receive radiation therapy once a day, five days a week for six weeks.

During treatment, patients will have a weekly exam, including blood work and urine tests. The blood work will include liver and kidney function tests as well as coagulation (blood clotting) tests.

Patients will be taken off study if intolerable side effects occur, including bleeding and/or severe allergic response.

During the 6 months after completion of radiation, while patients are still receiving rofecoxib, monthly medical histories, physical exams, blood tests, and urine tests will be performed. Patients will have a MRI at 1, 3, and 6 months after completion of radiation therapy.

The first year after completion of rofecoxib therapy, patients will be interviewed and examined with blood and urine tests and MRI every 3 months. During 1-3 years following completion of rofecoxib therapy, this will be repeated every 6 months. After 3 years following completion of rofecoxib, follow-ups will occur yearly.

This is an investigational study. Rofecoxib is currently approved by the FDA for use in adults only. A maximum of 30 patients will take part in this study at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed infiltrating lesion involving the pons and an MRI pattern of diffuse infiltration, that is not focal. The tumor may extend beyond the boundary of the pons.
* MRI of the brain with or without gadolinium within 4 weeks of starting therapy.
* Clinical history < 6 months duration
* Children >3 years of age and adults >18 years of age
* Treatment to begin within 6 weeks of diagnosis.
* Written informed consent
* Performance status: ECOG 0,1,2 or equivalent Lansky Play Performance Scale.
* All patients must have adequate bone marrow function (ANC>1000, platelets >100,000, SGPT < 2.5x ULN) and renal function (creatinine clearance >50/ml/min/1.73 m2 or age-adjusted serum creatinine < 3x ULN)

  * MRI of the spine within 4 weeks of starting therapy.

Exclusion Criteria:

* Pregnancy. All participants who are of child-bearing age must agree to use a method of birth control/pregnancy prevention.
* Bilirubin > 3x ULN.
* History of gastrointestinal bleeding.
* History of GI perforation due to ulcerative disease.
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Prior therapy (Dexamethasone is not considered therapy.)
* Prior malignancy
* Metastasis to the spine.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2001-10; Primary Completion 2004-10 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of VIOXX (rofecoxib) with 6 weeks of daily cranial radiation therapy | 1 month following radiation therapy
  Maximum Tolerated Dose defined using each level's dose limiting toxicity (DLT) and continuous reassessment method (CRM).

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Chang, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org